CLINICAL TRIAL: NCT02867774
Title: Impact of Physical Activity for Chronic Pelvic Pain
Acronym: IPA-CPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sara Till, MD, MPH, Minimally Invasive Gynecologic Surgery Fellow, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00112656
Record Dates: First submitted 2016-08-12; First posted 2016-08-16 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Pain
Keywords: chronic pelvic pain; central pain amplification; exercise; physical activity
MeSH Terms: conditions — Pelvic Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): This pilot study will enroll 25 women age 18-65 with greater than six months of noncyclic pelvic pain. Subjects will participate in an 8-week physical activity program specifically designed for patients with chronic pain and supervised by personal trainers and exercise physiologists in a rehab-focused, medically-based fitness center. Subjects will complete web-based assessment tools at the start of the program, immediately after completion of the 8-week program and four weeks after the conclusion of the program (at the 12-week time point).
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 8 week exercise program specifically designed for patients with chronic pain at Transitions Training Studio, a rehab-focused, medically-based fitness center based at the University of Michigan.
  The program is designed to gradually increase intensity and duration. If causes pain exacerbation, patients will go back to earlier level of intensity. It favors short, frequent activity episodes as this is often better tolerated than longer, infrequent episodes. The program begins with 30 minutes sessions 3 times per week with goal of increasing duration over course of the program.
  The program incorporates elements of flexibility, strength and cardio. Program design includes common elements but allows for a personalized program based on a subject's baseline fitness, interest and tolerance to activity. The program design emphasizes activities that patients can incorporate into their daily routine.

SUMMARY:
The purpose of this pilot study is to evaluate the impact of an intervention to increase physical activity on pain, function and quality of life in women with chronic pelvic pain.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to evaluate the impact of moderate-intensity physical activity on pelvic pain in women with chronic pelvic pain. We will develop a moderate-intensity physical activity program for patients with chronic pelvic pain in conjunction with exercise physiologists and physical medicine and rehabilitation (PM&R) physicians. Based on prior research in fibromyalgia and other centralized pain disorders, we hypothesize that eight weeks of moderate-intensity physical activity will reduce pain intensity and pain interference in women with chronic pelvic pain. We will also evaluate the impact of moderate-intensity physical activity on physical function, fatigue, sexual function, sleep, anxiety, depression, catastrophization and patient global impression of change in women with chronic pelvic pain. We hypothesize that eight weeks of moderate-intensity physical activity will result in improvements in these measures of function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-65 years old
* ≥ 6 months of noncyclic pelvic pain
* Pain that is severe enough to cause functional limitations, defined here as an average self-reported daily pain score of 4 on a 10 point scale
* Willing to attend activity session in Ann Arbor, MI at least 3 times per week
* English speaking

Exclusion Criteria:

* Pelvic surgery within the previous 3 months or plan for pelvic surgery within the following 3 months
* Participation in pelvic floor physical therapy during the 12 week study period
* Medical co-morbidities that prohibit participation in an exercise program, such as significant cardiovascular, pulmonary or orthopedic disease
* Pregnancy
* Documented history of significant dementia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Pain | 8 weeks
  Change in reported pain after physical activity intervention, measured using VAS and Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale

SECONDARY OUTCOMES:
Physical Function | 8 weeks
  Change in reported physical function, measured by the PROMIS Physical Function Scale
Fatigue | 8 weeks
  Change in reported fatigue, measured by the PROMIS Fatigue Scale
Sexual Function | 8 weeks
  Change in reported sexual function, measured by the Female Sexual Function Index
Sleep | 8 weeks
  Change in reported sleep, measured by the PROMIS Sleep Disturbance Scale
Anxiety | 8 weeks
  Change in reported anxiety, measured by the PROMIS Anxiety Scale
Depression | 8 weeks
  Change in reported depression, measured by the PROMIS Depression Scale
Catastrophization | 8 weeks
  Change in reported catastrophization, measured by the Pain Catastrophization Scale
Overall symptom improvement | 8 weeks
  Change in overall symptoms, measured by the Patient Global Impression of Change Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sawsan As-Sanie, MD, MPH, Principal Investigator — University of Michigan; Sara R Till, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Howard FM. Chronic pelvic pain. Obstet Gynecol. 2003 Mar;101(3):594-611. doi: 10.1016/s0029-7844(02)02723-0. PMID 12636968
- [Result] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Result] ACOG Committee on Practice Bulletins--Gynecology. ACOG Practice Bulletin No. 51. Chronic pelvic pain. Obstet Gynecol. 2004 Mar;103(3):589-605. No abstract available. PMID 14990428
- [Result] Williams DA, Clauw DJ. Understanding fibromyalgia: lessons from the broader pain research community. J Pain. 2009 Aug;10(8):777-91. doi: 10.1016/j.jpain.2009.06.001. PMID 19638325
- [Result] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Result] Tracey I, Bushnell MC. How neuroimaging studies have challenged us to rethink: is chronic pain a disease? J Pain. 2009 Nov;10(11):1113-20. doi: 10.1016/j.jpain.2009.09.001. PMID 19878862
- [Result] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Result] Brawn J, Morotti M, Zondervan KT, Becker CM, Vincent K. Central changes associated with chronic pelvic pain and endometriosis. Hum Reprod Update. 2014 Sep-Oct;20(5):737-47. doi: 10.1093/humupd/dmu025. Epub 2014 Jun 11. PMID 24920437
- [Result] As-Sanie S, Kim J, Schmidt-Wilcke T, Sundgren PC, Clauw DJ, Napadow V, Harris RE. Functional Connectivity is Associated With Altered Brain Chemistry in Women With Endometriosis-Associated Chronic Pelvic Pain. J Pain. 2016 Jan;17(1):1-13. doi: 10.1016/j.jpain.2015.09.008. Epub 2015 Oct 9. PMID 26456676
- [Result] As-Sanie S, Harris RE, Napadow V, Kim J, Neshewat G, Kairys A, Williams D, Clauw DJ, Schmidt-Wilcke T. Changes in regional gray matter volume in women with chronic pelvic pain: a voxel-based morphometry study. Pain. 2012 May;153(5):1006-1014. doi: 10.1016/j.pain.2012.01.032. Epub 2012 Mar 2. PMID 22387096
- [Result] As-Sanie S, Harris RE, Harte SE, Tu FF, Neshewat G, Clauw DJ. Increased pressure pain sensitivity in women with chronic pelvic pain. Obstet Gynecol. 2013 Nov;122(5):1047-1055. doi: 10.1097/AOG.0b013e3182a7e1f5. PMID 24104772
- [Result] Fontaine KR, Conn L, Clauw DJ. Effects of lifestyle physical activity on perceived symptoms and physical function in adults with fibromyalgia: results of a randomized trial. Arthritis Res Ther. 2010;12(2):R55. doi: 10.1186/ar2967. Epub 2010 Mar 30. PMID 20353551
- [Result] Fontaine KR, Conn L, Clauw DJ. Effects of lifestyle physical activity in adults with fibromyalgia: results at follow-up. J Clin Rheumatol. 2011 Mar;17(2):64-8. doi: 10.1097/RHU.0b013e31820e7ea7. PMID 21325963
- [Result] Larsson A, Palstam A, Lofgren M, Ernberg M, Bjersing J, Bileviciute-Ljungar I, Gerdle B, Kosek E, Mannerkorpi K. Resistance exercise improves muscle strength, health status and pain intensity in fibromyalgia--a randomized controlled trial. Arthritis Res Ther. 2015 Jun 18;17(1):161. doi: 10.1186/s13075-015-0679-1. PMID 26084281
- [Result] Busch AJ, Webber SC, Richards RS, Bidonde J, Schachter CL, Schafer LA, Danyliw A, Sawant A, Dal Bello-Haas V, Rader T, Overend TJ. Resistance exercise training for fibromyalgia. Cochrane Database Syst Rev. 2013 Dec 20;2013(12):CD010884. doi: 10.1002/14651858.CD010884. PMID 24362925
- [Result] Kayo AH, Peccin MS, Sanches CM, Trevisani VF. Effectiveness of physical activity in reducing pain in patients with fibromyalgia: a blinded randomized clinical trial. Rheumatol Int. 2012 Aug;32(8):2285-92. doi: 10.1007/s00296-011-1958-z. Epub 2011 May 19. PMID 21594719
- [Result] Soriano-Maldonado A, Ruiz JR, Aparicio VA, Estevez-Lopez F, Segura-Jimenez V, Alvarez-Gallardo IC, Carbonell-Baeza A, Delgado-Fernandez M, Ortega FB. Association of Physical Fitness With Pain in Women With Fibromyalgia: The al-Andalus Project. Arthritis Care Res (Hoboken). 2015 Nov;67(11):1561-70. doi: 10.1002/acr.22610. PMID 25939406
- [Result] Johannesson E, Simren M, Strid H, Bajor A, Sadik R. Physical activity improves symptoms in irritable bowel syndrome: a randomized controlled trial. Am J Gastroenterol. 2011 May;106(5):915-22. doi: 10.1038/ajg.2010.480. Epub 2011 Jan 4. PMID 21206488
- [Result] Johannesson E, Ringstrom G, Abrahamsson H, Sadik R. Intervention to increase physical activity in irritable bowel syndrome shows long-term positive effects. World J Gastroenterol. 2015 Jan 14;21(2):600-8. doi: 10.3748/wjg.v21.i2.600. PMID 25593485
- [Result] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Result] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2015 Jan 9;1(1):CD004376. doi: 10.1002/14651858.CD004376.pub3. PMID 25569281
- [Result] Fransen M, McConnell S, Hernandez-Molina G, Reichenbach S. Exercise for osteoarthritis of the hip. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD007912. doi: 10.1002/14651858.CD007912.pub2. PMID 24756895
- [Result] Santiago MD, Carvalho Dde S, Gabbai AA, Pinto MM, Moutran AR, Villa TR. Amitriptyline and aerobic exercise or amitriptyline alone in the treatment of chronic migraine: a randomized comparative study. Arq Neuropsiquiatr. 2014 Nov;72(11):851-5. doi: 10.1590/0004-282x20140148. PMID 25410451
- [Result] Ortiz MI, Cortes-Marquez SK, Romero-Quezada LC, Murguia-Canovas G, Jaramillo-Diaz AP. Effect of a physiotherapy program in women with primary dysmenorrhea. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:24-9. doi: 10.1016/j.ejogrb.2015.08.008. Epub 2015 Aug 17. PMID 26319652
- [Result] Ozdemir S, Bebis H, Ortabag T, Acikel C. Evaluation of the efficacy of an exercise program for pregnant women with low back and pelvic pain: a prospective randomized controlled trial. J Adv Nurs. 2015 Aug;71(8):1926-39. doi: 10.1111/jan.12659. Epub 2015 Mar 31. PMID 25823561
- [Result] Gavi MB, Vassalo DV, Amaral FT, Macedo DC, Gava PL, Dantas EM, Valim V. Strengthening exercises improve symptoms and quality of life but do not change autonomic modulation in fibromyalgia: a randomized clinical trial. PLoS One. 2014 Mar 20;9(3):e90767. doi: 10.1371/journal.pone.0090767. eCollection 2014. PMID 24651512
- [Result] Hooten MW, Qu W, Townsend CO, Judd JW. Effects of strength vs aerobic exercise on pain severity in adults with fibromyalgia: a randomized equivalence trial. Pain. 2012 Apr;153(4):915-923. doi: 10.1016/j.pain.2012.01.020. Epub 2012 Feb 15. PMID 22341565
- [Result] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Result] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359